CLINICAL TRIAL: NCT00667212
Title: Individual Cognitive Behavioral Psychotherapy for Intermittent Explosive Disorder
Brief Title: Psychotherapy for Intermittent Explosive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 15143A
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Anger; Intermittent Explosive Disorder
Keywords: anger; intermittent; explosive
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders | interventions — Cognitive Behavioral Therapy; Cognitive Restructuring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Supportive Psychotherapy
  Interventions: Behavioral: Supportive Psychotherapy
- 1 (Active Comparator): Cognitive Behavioral Therapy (Cognitive Restructuring, Relaxation, and Coping Skills Training: CRCST)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Twelve weekly therapy sessions, approximately one hour each in duration
  Other Names: Cognitive Restructuring, Relaxation, and Coping Skills Training
  Arms: 1
Behavioral: Supportive Psychotherapy — Twelve weekly therapy sessions, approximately one hour each in duration
  Arms: 2

SUMMARY:
The goal of this study is to examine the effectiveness two forms of psychotherapy (also known as "talk therapy" ) for individuals with anger and aggression problems. Anger and aggression are everywhere - on the road, in the schools, at little league games, at home, and at work. In this study we are testing usefulness of anger management techniques in reducing symptoms of Intermittent Explosive Disorder (IED) and impulsive, aggressive behavior.

DETAILED DESCRIPTION:
Qualified participants will be randomly assigned to 12 1-hour sessions of either cognitive-behavioral therapy or supportive psychotherapy.

Participation in this study will require 13 visits over approximately 4 months with a 3 follow-up session. Therapy is provided at no cost and each study participant will receive a comprehensive psychological assessment. Two types of talk therapy are being offered in this study. One form of therapy focuses on thought and behaviors associated with anger and aggression. This type of therapy is known as cognitive behavioral therapy. The other type of therapy focuses on the individuals' feeling about their anger /aggression and the situations that lead to this anger. This is known as supportive therapy. The form of therapy you are given will be randomly determined (like by flipping of a coin).

ELIGIBILITY:
Inclusion Criteria:

* Have problems with anger, temper outbursts, being irritable, getting in trouble at work or at home because of impulsive/aggressive behavior.
* Between the ages of 18 and 55.
* Meet other eligibility requirements as outlined by the research protocol.

Exclusion Criteria:

* Lifetime diagnosis of psychosis or bipolar disorder
* Current diagnosis of substance dependence or major depressive disorder.
* Current suicidal or homicidal ideation,
* Recent use of selective serotonin reuptake inhibitors (past month) or other psychotropic medication (past two months)
* Recent psychotherapy for aggression (past six months.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in Overt Aggression Scale - Modified (OASM) Score | Up to 12 months
  Items are scored on a 5-point scale. Higher scores indicate higher levels of aggression.
Change in State-Trait Anger Expression Inventory - Trait Anger Scale [STAXI-2] | Up to 12 months
  Items are scored on a 4-point scale. Higher scores indicate high levels of anger.
Change in Hostile Automatic Thoughts (HAT) Scale | Up to 12 months
  Each item is answered on a 5-point Likert scale ranging from 0=not at all to 5=all the time. Higher scores indicate higher frequency of hostile thoughts experienced.

SECONDARY OUTCOMES:
Change in Self-Report of Aggression and Social Behavior Measure (SRASBM) Score | Up to 12 months
  Items are scored on a 7-point scale to indicate how truthfully the statement describes personal experiences during the past year, ranging from 0=not at all true to 7=very true. Higher scores indicate high levels of aggression
Change in Social Information Processing-Attribution and Emotional Response Questionnaire (SIP-AEQ) Score | Up to 12 months
  Items are scored on a 0-3 Likert scale (0 = not at all likely to 3 = extremely likely). Higher scores indicate higher levels of hostility.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McCloskey, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States